CLINICAL TRIAL: NCT04469985
Title: Allogeneic Stem Cell Transplantation (ALLO-SCT) in Elderly: 17-years Retrospective GITMO Survey
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Prof Domenico Russo, PI, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: GITMO-AlloElderly
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Allogeneic Stem Cell Transplantation in Elderly Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The age of patients' population is increasing every year, as the life expectancy. Thus, the incidence and prevalence of hematological cancers is increasing. In particular, acute leukemias and myelodisplastic syndromes are the most frequent diseases of the hematopoietic system. Allogeneic stem cell transplantation (allo-SCT) is the main therapeutic options for these diseases, and the number of allo-SCTs in the elderly is currently in progressive growth. This is partially due to the improvement of the allo-SCT procedure over the years, with the amelioration of donor selection, HLA typing, graft versus host disease (GVHD) and infections prophylaxis and treatment.

Nevertheless, there is still an unmet clinical need, represented by the lack of extensively and detailed outcome analysis of elderly patients addressed to allo-SCT. With this aim, we planned this retrospective analysis of allo-SCTs in patients older than 60 years, within the GITMO transplant activity of the last 17 years. This study will help us in designing future prospective trials, including a comprehensive geriatric assessment of frailty, in order to address to allo-SCT those elderly who have the highest probability to achieve the best long term outcome with the lowest transplant-related mortality and morbidity.

ELIGIBILITY:
This study will enrol patients older than 60 years who received hematopoietic stem cell transplantation (HSCT) between 1st January 2000 and 31st December 2017.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enrol patients older than 60 years who received hematopoietic stem cell transplantation (HSCT) between 1st January 2000 and 31st December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 2061 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  Overall Survival
Disease Free Survival | 1 year
  Disease Free Survival
Transplant Related Mortality | 1 year
  Transplant Related Mortality
Acute Graft Versus Host Disease Incidence | 100 days
  Acute Graft Versus Host Disease Incidence
Chronic Graft Versus Host Disease Incidence | 1 year
  Chronic Graft Versus Host Disease Incidence
Relapse Incidence | 1 year
  Relapse Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Michele Malagola, MD, Principal Investigator — Bone Marrow Transplant Unit, University of Brescia
Locations (1):
- Chair of Hematology and Bone marrow Transplant Unit, Brescia, Italy

REFERENCES:
- [Derived] Malagola M, Polverelli N, Rubini V, Martino M, Patriarca F, Bruno B, Giaccone L, Grillo G, Bramanti S, Bernasconi P, De Gobbi M, Natale A, Terruzzi E, Olivieri A, Chiusolo P, Carella AM, Casini M, Nozzoli C, Mazza P, Bassi S, Onida F, Vacca A, Falcioni S, Luppi M, Iori AP, Pavone V, Skert C, Carluccio P, Borghero C, Proia A, Selleri C, Sacchi N, Mammoliti S, Oldani E, Ciceri F, Russo D, Bonifazi F. GITMO Registry Study on Allogeneic Transplantation in Patients Aged >/=60 Years from 2000 to 2017: Improvements and Criticisms. Transplant Cell Ther. 2022 Feb;28(2):96.e1-96.e11. doi: 10.1016/j.jtct.2021.11.006. Epub 2021 Nov 21. PMID 34818581